CLINICAL TRIAL: NCT00397228
Title: Optimizing the Performance of ALTROPANE® SPECT Imaging in Patients With Parkinson Disease
Brief Title: ALTROPANE® SPECT Imaging in Patients With Parkinson Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, Principal Investigator, Molecular NeuroImaging
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALTROPANE dosing
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson; imaging; dopamine transporter
MeSH Terms: conditions — Parkinson Disease | interventions — N-iodoallyl-2-carbomethoxy-3-(4-fluorophenyl)tropane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALTROPANE® (Experimental): ALTROPANE® dosing
  Interventions: Drug: ALTROPANE®

INTERVENTIONS:
Drug: ALTROPANE® — ALTROPANE® SPECT imaging

SUMMARY:
After a screening evaluation including baseline clinical laboratory testing, a physical and neurological evaluation, subjects will be asked to undergo an injection of ALTROPANE® followed by up to 60 minutes of serial dynamic imaging. Subjects will undergo a second injection of ALTROPANE® followed by up to 60 minutes of serial dynamic imaging within 2-6 weeks of the injection 1.

DETAILED DESCRIPTION:
The underlying goal of this open label imaging study is to optimize the imaging outcome for ALTROPANE® in mild to moderate PD subjects. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Subjects with PD (n=15) will be recruited to undergo ALTROPANE® SPECT. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a physical and neurological evaluation. Subjects will be asked to undergo an injection of ALTROPANE® followed by up to 60 minutes of serial dynamic imaging. Subjects will be asked to undergo a second imaging visit two-six weeks following the initial imaging visit to assess the reproducibility of the imaging outcome. The imaging analyses will be performed by an image-processing specialist who will remain masked to clinical severity. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a target region to occipital ratio. Striatal regions of interests for caudate and putamen will be defined and placement standardized based on previously optimized region placement protocols. Imaging data will also be analyzed using an automated objective striatal analysis software package.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 30 years or older at time of PD diagnosis.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of idiopathic Parkinson's disease of < 7 years.
* Hoehn and Yahr stages I-III.
* Negative drug screen

Exclusion Criteria:

* The participant has atypical or drug-induced Parkinson's disease.
* The participant has dementia.
* The participant has a clinically significant clinical laboratory value and/or clinically significant unstable medical or psychiatric illness.
* Treatment within the six months prior to screening with bupropion, methylphenidate, reserpine, alpha methyldopa, or amphetamine.
* The participant has a history of alcohol, narcotic, or any other drug abuse within the past 2 years.
* The participant has received an investigational drug within 60 days of screening visit.
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Optimize ALTROPANE® dosing and the image acquisition protocol to develop a quantitative imaging outcome that would enhance ALTROPANE® reliability, ease of use and ease of analysis. | 2 years

SECONDARY OUTCOMES:
Evaluate a state-of-art automated objective striatal analysis tool for ALTROPANE® and to test the reliability of these quantitative outcomes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Molecular NeuroImaging
Locations (1):
- Molecular NeuroImaging, New Haven, Connecticut, United States